CLINICAL TRIAL: NCT04346524
Title: SweMaMi DM1, Diabetic Women's Microbiome During Pregnancy
Brief Title: SweMaMi DMI, Microbiome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Wiberg-Itzel, Associate professor, Karolinska Institutet
Other Study IDs: DM1
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Microbioma; maternal and fetal pregnacy outcomes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- microbiome sampling: pregnant women with type 1 diabetes
  Interventions: Other: sampling of microbiome

INTERVENTIONS:
Other: sampling of microbiome — women will sample from vagina, feces, and saliva during pregnancy

SUMMARY:
Dysbiosis is associated with an increased risk of preeclampsia during pregnancy. The microbiome differs between those with and without type 1 diabetes and the cause of type 1 diabetes has been associated with dysbiosis. Increased knowledge of the microbiome and its variation, depending on the state of health during pregnancies complicated with type 1 diabetes, could in the future lead to preventive care and treatments during these pregnancies.

DETAILED DESCRIPTION:
Prospective cohort. All women with type 1 diabetes that are planning a pregnancy and being cared for at the diabetic ward at Södersjukhuset will be asked to participate, n= 55.

All pregnancies complicated with type 1 diabetes that are being cared for at the special maternity ward at Södersjukhuset, n=45.

The expected to include is 100. Expected viable pregnancies: 50.

The maternal vaginal, fecal and oral microbiome will be sampled by "self-sampling" at home before, during and after the pregnancy, by this schedule:

1. Inclusion, before pregnancy after an appointment with the diabetic doctor or nurse. Or at the first visit at the special maternity care ward during pregnancy (around gestational week 8).
2. When the pregnancy is first discovered if the inclusion were before pregnancy.
3. Week 28.
4. When attending delivery ward in labor
5. 6-10 weeks postpartum from both the mother and the new-born. The tests will be sent to the obstetric research center at Södersjukhuset, where the tests will be saved in freezes. The analysis will be performed at CTMR at the Karolinska Institute.

Background, pregnancy and delivery data will then be associated with the woman microbiome in the vagina, in feces and in saliva.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women with type 1 diabetes
* Included as a patient at women's clinic Soderhospital in Stockholm
* Acceptant to sample her microbiome during pregnancy

Exclusion Criteria:

* Women without type 1 diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women with type 1 diabetes
Study Population: pregnant women with type 1 diabetes
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Maternal complications during pregnancy | through study completion, an average of 1 year
  The frequency of Preeklampsia, hypertension and other pregnancy complications

SECONDARY OUTCOMES:
Fetal complications during pregnancy | through study completion, an average of 1 year
  Large for gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Eva Wiberg-Itzel, PhD, Principal Investigator — Karolinska Institute Sodersjukhuset Sweden
Locations (2):
- Sweden (2):
  - Eva Wiberg-Itzel, Danderyd, Sverige
  - Eva Wiberg-Itzel, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided
We have not discussed this question yet